CLINICAL TRIAL: NCT01397721
Title: Pulmonary Vascular Changes in Early Chronic Obstructive Pulmonary (MESA-COPD)
Brief Title: Pulmonary Vascular Changes in Early Chronic Obstructive Pulmonary
Acronym: MESA-COPD
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, R. Graham Barr, Irving Associate Professor of Medicine and Associate Professor of Epidemiology, Columbia University
Other Study IDs: AAAD6395; R01HL093081-01 (NIH)
Record Dates: First submitted 2011-07-13; First posted 2011-07-20 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD); pulmonary vasculature; pulmonary hypertension; atherosclerosis; smokers; emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary; Atherosclerosis; Emphysema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be stored at Columbia and at University of Vermont, identified only by study ID and following standard procedures. It will be accessible only to study investigators and, if the participant approves, outside investigators following MESA/NIH protocols and with IRB approval. Blood will be kept indefinitely.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Multi-Ethnic Study of Atherosclerosis (MESA) - Chronic Obstructive Pulmonary Disease (COPD) Study aims to characterize the pulmonary vascular changes and their biology in early COPD using imaging, gene expression profiling and peripheral cellular measures.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is the third leading cause of death in the US and will soon replace stroke as the third leading cause.

Translation of promising biological hypotheses of COPD pathogenesis to human populations that may lead to new therapies is urgently needed. The vascular hypothesis of COPD was articulated almost 50 years ago. Bench research on endothelial dysfunction in COPD is evolving rapidly and has shown that acrolein in cigarette smoke causes endothelial apoptosis and endothelial apoptosis is directly implicated in COPD pathogenesis. Clinical studies on endothelial dysfunction and vascular changes in COPD are limited.

The proposed study is a longitudinal study of smokers nested among the MESA-Lung (AAAA7791) and EMphysema and Cancer Action Project (EMCAP) Studies (AAAA6484), which together provide a well-defined cohort of 4,617 participants with prior spirometry and CT measures.

The Multiethnic Study of Atherosclerosis - Chronic Obstructive Pulmonary Disease (MESA COPD Study) has two main scientific purposes:

1. characterize the pulmonary vascular changes in COPD and their biology, and
2. propose novel pathways for new therapies in COPD.

MESA COPD is a longitudinal study of smokers nested within the MESA-Lung and EMCAP cohorts of 360 participants (160 cases with mild, 60 cases with moderate and 40 cases with severe COPD and 100 controls) who will be phenotyped with magnetic resonance (MR) pulmonary angiography, pulmonary function testing, full-lung CT scans, serum Vascular Endothelial Growth Factor (VEGF), cell assays and gene expression profiling. MESA COPD Study will contribute improving the knowledge of early changes in COPD that may lead to novel disease-modifying medical therapies and preventative strategies.

ELIGIBILITY:
Inclusion Criteria:

* age 50-79 years at time of enrollment
* ever smokers (10 or more pack-years)
* participation in MESA or EMCAP studies

Exclusion Criteria:

* clinical cardiovascular disease (left congestive heart failure (CHF), valve disease, coronary artery disease (CAD), stroke, or congenital heart disease),
* asthma, pulmonary embolism or lung disease other than COPD,
* weight > 300 lbs,
* chronic renal insufficiency ([estimated glomerular filtration rate (eGFR)] < 45 mL/min/1.73 m2),
* atrial fibrillation, and
* contraindications to magnetic resonance imagine (MRI), gadolinium, albuterol or spirometry testing.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately Study Subjects:
  MESA COPD will recruit approximately 360 participants from EMCAP at Columbia, and from MESA at Columbia; JH University; North Western University; and University of California.
  Cases will be defined according to the current American Thoracic Society/European Respiratory Society (ATS/ERS) definition of COPD of a post-bronchodilator capacity (FEV1/FVC) ratio < 0.70 and classified as mild, moderate and severe as post-bronchodilator FEV1 of 80-100% predicted, 50-80% predicted and < 50% predicted, respectively.
  Controls will be defined in the above sampling frame as those with normal lung function (pre-bronchodilator FEV1/FVC ratio >= 0.70, and no restrictive ventilatory defect.
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in cardiac structure and pulmonary vascular structure and function | Up to 2 years from start of study
  Cardiac structure: changes in right ventricular (RV) mass, RV mass/Right Ventricular End-Diastolic Volume (RV-EDV)
  Pulmonary structure: changes in total pulmonary vascular volume (TPVV) and pulmonary artery (PA) perfusion
  Function: changes in PA flow and distensibility

SECONDARY OUTCOMES:
Number of CD31+/CD42 endothelial microparticles (EMPs) | Up to 2 years from the start of study
  Numbers of CD31+/CD42 EMPs reflective of apoptosis are elevated; They are abnormal in severe, moderate and mild COPD compared to controls.
Number of circulating endothelial cells (CEC) | Up to 2 years from the start of study
  Numbers of circulating endothelial cells (CEC), resulting from endothelial injury, are elevated. They are abnormal in severe, moderate and mild COPD compared to controls
Number of endothelial progenitor cells (EPCs), involved in endothelial repair, are decreased | Up to 2 years from the start of study
  They are abnormal in severe, moderate and mild COPD compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: R. Graham Barr, MD, DrPh, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - UCLA Research Center, Alhambra, California
  - Northwestern University Medical School, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University, New York, New York

REFERENCES:
- See also: Related Info — http://www.mesa-nhlbi.org/